CLINICAL TRIAL: NCT00967902
Title: The REMEDEE Study: A Prospective, Randomized Study to Evaluate the Safety and Efficacy of an Abluminal Sirolimus Coated Bio-engineered Stent (Combo Bio-engineered Sirolimus Eluting Stent)
Brief Title: Safety and Effectiveness Study of Combo Bio-engineered Sirolimus Eluting Stent
Acronym: REMEDEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OrbusNeich (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VP-0427
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Lesions
Keywords: intracoronary stent; drug eluting stent; sirolimus; endothelial progenitor cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combo (Experimental): The Combo Stent is composed of the OrbusNeich R stent™, with an abluminal coating of a bioabsorbable polymer matrix formulated with sirolimus for sustained release, and an anti-CD34 antibody cell capture coating on the luminal surface.
  Interventions: Device: coronary stenting
- Taxus® Liberté® Stent (Active Comparator): Commercially available product
  Interventions: Device: coronary stenting

INTERVENTIONS:
Device: coronary stenting — Balloon dilatation of obstructive coronary artery disease with deployment of a metallic stent to scaffold the dilated lesion; stent incorporating sustained release of anti-proliferative agent to control neointimal proliferation and reocclusion; test device incorporates affinity surface for circulating EPCs

SUMMARY:
To demonstrate the safety and effectiveness of the Combo Bio-engineered Sirolimus Eluting Stent (Combo Stent) compared to the Taxus® Liberté® Stent in the treatment of coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* The patient must be ≥18 and ≤ 80 years of age;
* Symptomatic ischemic heart disease (CCS class 1-4, Braunwald Class IB, IC, IIB, IIC, IIIB, IIIC, and/or objective evidence of myocardial ischemia);
* Acceptable candidate for CABG;
* The Patient is willing to comply with specified follow-up evaluations;
* The Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics Committee (MEC), Institutional Review Board (IRB), or Human Research Ethics Committee (HREC).

Angiographic Inclusion Criteria:

* Single de novo or non-stented restenotic lesion in the target vessel;
* Patients with two-vessel coronary disease, may have undergone successful treatment (<20% diameter stenosis by visual estimate) of the non-target vessel with approved devices up to and including the index procedure but must be prior to the index target vessel treatment. Any non-target vessel or lesion intended to be treated during the index procedure, cannot be an unprotected left main, ostial lesion, chronic total occlusion (CTO), heavily calcified, bifurcation, vein grafts, have angiographic evidence of thrombus, be anything requiring atherectomy, thrombectomy, or pre-treatment with anything other than balloon angioplasty;
* Target lesion located in a native coronary artery;
* Target lesion (maximum length is 20 mm by visual estimate) covered by a single stent maximum 23 mm length for Combo Stent, and 24 mm in length for TAXUS® Liberté® (stent coverage including at least 3 mm of healthy vessel is recommended). The lesion length should be measured after pre-dilation procedure;
* Reference vessel diameter must be ≥2.5 to ≤ 3.5 mm by visual estimate. The vessel diameter should be measured after pre-dilation procedure and after intra-coronary nitroglycerin if spasm is suspected;
* Target lesion ≥50% and <100% stenosed by visual estimate.

Exclusion Criteria:

General Exclusion Criteria:

* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test;
* Patient has had a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure (elevated troponin or CK-MB ≥2 times upper limit of normal) or >72 hours preceding the index procedure and CK and CK-MB have not returned to within normal limits at the time of procedure;
* The patient is currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate unresponsive prolonged chest pain;
* Impaired renal function (serum creatinine >2.0 mg/dL or 177 μmol/l) or on dialysis;
* Platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a WBC <3,000 cells/mm3;
* Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated;
* Patient requires low molecular weight heparin (LMWH) treatment post-procedure or has received a dose of LMWH ≤8 hours prior to index procedure;
* Patient has received any organ transplant or is on a waiting list for any organ transplant;
* Patient has other medical illness (e.g., cancer, known malignancy, or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year);
* Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, prasugrel, stainless steel alloy, sirolimus, paclitaxel and/or contrast sensitivity that cannot be adequately pre-medicated;
* Patient has previously received murine therapeutic antibodies and exhibited sensitization through the production of Human Anti-Murine Antibodies (HAMA);
* Patient presents with cardiogenic shock;
* Patient has current unstable cardiac arrhythmias that create hemodynamic instability;
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion;
* Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
* Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up;

Angiographic Exclusion Criteria:

* Unprotected left main coronary artery disease with ≥50% stenosis;
* Ostial target lesion(s);
* Totally occluded target vessel (TIMI flow 0);
* Calcified target lesion(s) which cannot be successfully predilated;
* Target lesion has excessive tortuosity unsuitable for stent delivery and deployment;
* Angiographic evidence of thrombus in the target lesion(s);
* Target lesion involving bifurcation with a side branch ≥2.0 mm in diameter (either stenosis of both main vessel and major side branch or stenosis of just major side branch) that would require intervention of diseased side branch;
* A significant (>50%) stenosis proximal or distal to the target lesion that cannot be covered by same single stent;
* Diffuse distal disease to target lesion with impaired runoff;
* Left ventricular ejection fraction (LVEF) ≤30% (LVEF must be obtained within 6 months prior to the index procedure);
* Pre-treatment with devices other than balloon angioplasty;
* Prior stent within 10 mm of target lesion;
* Intervention (PCI or bypass) of another lesion performed within 6 months before or planned within 30 days following the index procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss of the Combo Stent compared to the TAXUS® Liberté® DES | 9 months post-procedure.

SECONDARY OUTCOMES:
All-cause and cardiac mortality | 30 days, 9 months, 1, 2, 3, 4, and 5 year
Myocardial infarction: Q-wave and non Q-wave, cumulative and individual | 30 days, 9 months, 1, 2, 3, 4, and 5 years
Major Adverse Cardiac Event (MACE) defined as a composite of death, MI (Q-wave or non Q-wave), emergent CABG, or target lesion revascularization by repeat PTCA or CABG | Hospital discharge, 30 days, 9 months, 1, 2, 3, 4 and 5 years post-procedure
Vascular complications from index procedure | Up to hospital discharge
Rate of stent thrombosis, per ARC definition of definite and probable stent thrombosis further categorized as early, late or very late | 30 days, 9 months, 1, 2, 3, 4 and 5 years post-procedure
Change in human anti-murine antibody (HAMA) plasma levels | 30 day and 9 month follow-up compared to baseline
Device success, defined as attainment of <50% residual stenosis of the target lesion using the Combo Stent | Index procedure
Lesion success defined as attainment of < 50% residual stenosis using any percutaneous method | Index procedure
Procedure success defined as lesion success without the occurrence of in-hospital MACE | Up to hospital discharge
Clinically (ischemia)-driven target lesion revascularization | 30 days, 9 months, 1, 2, 3, 4 and 5 years
Clinically (ischemia)-driven target vessel revascularization | 30 days, 9 months, 1, 2, 3, 4 and 5 years
In-stent and in-segment angiographic binary restenosis | 9 months
In-stent and in-segment minimum lumen diameter (MLD) | 9 months
In-stent, proximal and distal late lumen loss | 9 months
Neointimal hyperplasia volume and % in-stent volume obstruction as measured by intravascular ultrasound (IVUS) for patients receiving angiographic/IVUS follow-up | 9 months
Target lesion failure (TLF) (defined as death, MI and ischemic target lesion revascularization (TLR)) | 30 days, 9 months, 1, 2, 3, 4 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian T Meredith, MBBS, PhD, Principal Investigator — Monash University; Stephan Windecker, MD, Principal Investigator — University of Bern; Alexandre Abizaid, MD, Principal Investigator — Inst Dante Pazzanese of Cardiology; Roxana Mehran, MD, Study Director — CardioVascular Research Foundation; Alexandra Lansky, MD, Study Director — CardioVascular Research Foundation
Locations (1):
- John Hunter Hospital, Newcastle, New South Wales, Australia

REFERENCES:
- [Result] Haude M, Lee SW, Worthley SG, Silber S, Verheye S, Erbs S, Rosli MA, Botelho R, Meredith I, Sim KH, Stella PR, Tan HC, Whitbourn R, Thambar S, Abizaid A, Koh TH, Den Heijer P, Parise H, Cristea E, Maehara A, Mehran R. The REMEDEE trial: a randomized comparison of a combination sirolimus-eluting endothelial progenitor cell capture stent with a paclitaxel-eluting stent. JACC Cardiovasc Interv. 2013 Apr;6(4):334-43. doi: 10.1016/j.jcin.2012.10.018. Epub 2013 Mar 20. PMID 23523459